CLINICAL TRIAL: NCT01017913
Title: Effects of Transcutaneous Electrical Nerve Stimulation (TENS) and Interferential Currents (IFC) in Patients With Non Specific Chronic Low Back Pain: Randomized Clinical Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation and Interferential Currents in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Centro Universitario de Maringa (Other)
Responsible Party: Effects of Transcutaneous Electrical Nerve Stimulation (TENS) and Interferential Currents (IFC) in patients with non specific chronic low back pain: randomized clinical trial, Unifesp/ Cesumar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0143/06
Record Dates: First submitted 2009-09-22; First posted 2009-11-23 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Low Back Pain
Keywords: rehabilitation; electrotherapy; back pain
MeSH Terms: conditions — Back Pain | interventions — Transcutaneous Electric Nerve Stimulation; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Electrotherapy equipment (Active Comparator): The TENS equipment was calibrated on 20 hertz frequency, and a pulse width of 330 ms with two channels.
  Interventions: Other: TENS; Other: Interferential currents
- electrotherapy equipment (Active Comparator): The CI was adjusted with 4000 HZ bases frequency, modulation frequency range 20 HZ, ∆F10 HZ, slope 1/1 and quadripolar manner.
  Interventions: Other: TENS; Other: Interferential currents
- Control (No Intervention): The patients of the Control group stayed without any treatment in the same period
  Interventions: Other: TENS

INTERVENTIONS:
Other: TENS — The TENS equipment was calibrated on 20 hertz frequency, and a pulse width of 330 ms (standing in control number seven) with two channels.
  Other Names: Transcutaneous electrical nervous stimulation
Other: Interferential currents — The IFC was adjusted to a base frequency of 4000 Hz, with a modulation frequency range of 20 Hz, ∆F of 10 Hz and slope of 1/1, in quadripolar mode.
  Other Names: IFC: intereferential currents; electrotherapy
  Arms: Electrotherapy equipment; electrotherapy equipment

SUMMARY:
The purpose of this study was to compare the effects of the TENS and IFC in patients with non specific chronic low back pain.

DETAILED DESCRIPTION:
Setting Outpatient physiotherapy department in university (Cesumar)

Participants A hundred and fifty patients with non specific chronic low back pain with or without radicular pain.

Interventions The patients were randomly divided into three groups: 1) TENS; 2) IFC; e 3) Control. Ten sessions of electrotherapy for groups 1 and 2, while the patients of the Control group stayed without any treatment in the same period

Main Outcome Measures Intensity of the pain through the Visual Analogue Scale and McGill Pain Questionnaire; specific functional disability by Roland Morris Disability Questionnaire; Analgesic period (hours); and the medication consumption

Statistic Analysis All data were analyzed using Statistica version 7 and SAS version 9.1. Baseline characteristics were compared using the Shapiro-Wilks test for continuous variables and then analysis of variance for measuring independent data. The characteristics of the patients who finished the treatment were compared with those of the lost patients, using one-way ANOVA and the Kruskal-Wallis test.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who had had low back pain for less than three months

Exclusion Criteria:

* Individuals who were receiving treatment for their pain with another method at the same time, except for medicines;
* Pregnant women;
* Patients who had undergone vertebral column surgery (less than three months before the time of this study);
* Individuals with contraindications against electrotherapy, such as skin lesions, abnormal sensitivity, infectious and blood diseases, heart pacemakers or inability to answer questionnaires;
* Patients with fibromyalgia;
* Individuals with psychiatric problems;
* Individuals who refused to participate or were unwilling to follow a protocol lasting for two weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pain and Disability | Before and after ten sessions (interventions groups) or ten days (control group)

SECONDARY OUTCOMES:
Analgesic period (hours)and medication consumption | before and after ten sessions (interventions groups) or ten days (control group)

CONTACTS AND LOCATIONS:
Overall Officials: Ligia M Facci, Principal Investigator — Unifesp/ Cesumar
Locations (1):
- Cesumar, Maringá, Paraná, Brazil

REFERENCES:
- [Derived] Facci LM, Nowotny JP, Tormem F, Trevisani VF. Effects of transcutaneous electrical nerve stimulation (TENS) and interferential currents (IFC) in patients with nonspecific chronic low back pain: randomized clinical trial. Sao Paulo Med J. 2011;129(4):206-16. doi: 10.1590/s1516-31802011000400003. PMID 21971895